CLINICAL TRIAL: NCT00076557
Title: A Phase I Safety Study in Subjects With Severe Hemophilia B (Factor IX Deficiency) Using Adeno-Associated Viral Vector to Deliver the Gene for Human Factor IX Into the Liver
Brief Title: Safety of a New Type of Treatment Called Gene Transfer for the Treatment of Severe Hemophilia B
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avigen (Industry)
Collaborators: Stanford University (Other); Children's Hospital of Philadelphia (Other); The Hemophilia Center of Western Pennsylvania (Other); University of Washington (Other); The University of Texas Health Science Center, Houston (Other); University of Campinas, Brazil (Other); Christian Medical College, Vellore, India (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB IND 9398
Record Dates: First submitted 2004-01-26; First posted 2004-01-28 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2004-01

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; Factor IX; Gene Transfer; Adeno-Associated Virus (AAV)
MeSH Terms: conditions — Hemophilia B

INTERVENTIONS:
Genetic: Adeno-Associated Viral with Human Factor IX

SUMMARY:
In this study a modified virus called adeno-associated virus (AAV) will be used to transfer a normal gene for human clotting factor IX into patients with severe hemophilia B (AAV human Factor IX vector). Gene therapy is a very new medical technique being used in a number of clinical studies for diseases such as cancer and cystic fibrosis. At this time, the U.S. Food and Drug Administration has approved no gene transfer products for commercial use. To date, 8 subjects have received AAV vector in the muscle for a hemophilia B trial by intramuscular injection, and, to date, 6 subjects have been treated with AAV vector in the current hemophilia B liver trial. Eleven cystic fibrosis subjects have received AAV vector into their nasal sinuses or lungs to date. In this study, AAV human Factor IX vector will be injected into the liver using a catheter inserted into a large blood vessel (called the proper hepatic artery or the right hepatic artery).

ELIGIBILITY:
* Males with severe hemophilia B with Factor IX activity level < 1% of normal.
* Life expectancy of > 1 year.
* Age > 18 years old.
* Ability to give informed consent.
* Greater than twenty exposure days of treatment with Factor IX protein.
* No history or presence of an inhibitor to Factor IX protein.
* Subjects must be able to receive Factor IX protein on a home infusion protocol.
* Subjects must have a normal protime (PT).
* Hepatitis C infected subjects will be evaluated for liver fibrosis based on liver biopsy data graded on a scale of 0-4 (Poynard et. al., 1997). Subjects who are Hepatitis C antibody and RNA positive and have not had a liver biopsy within the last 36 months will be required to have one.
* Subjects must have low AAV titer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-01

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Avigen Ongoing Clinical Trials — http://www.avigen.com/research.php